CLINICAL TRIAL: NCT06727747
Title: Effect of Cervical Traction on Balance Parameters in Patients with Cervical Radiculopathy: a Randomized Controlled Trial
Brief Title: Effect of Cervical Traction on Balance in Cervical Radiculopathy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Monastir (Other)
Responsible Party: Principal Investigator, Anis Jellad, Professor, University of Monastir
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CTRB
Record Dates: First submitted 2024-10-14; First posted 2024-12-11 (Actual); Last update posted 2024-12-11 (Actual); Status verified 2024-12

CONDITIONS: Cervical Radiculopathy; Balance Disorders
MeSH Terms: conditions — Radiculopathy | interventions — Rehabilitation

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: The clinician who screened patients for eligibility
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Group A (Sham Comparator): Patients in group A recieved cervical traction with 2 kg load combined with standard rehabilitation program. This group is condidered as sham because the 2 kg load does not have any effect on anatomical structures of the cervical spine.
  Interventions: Other: Cervical traction; Other: Rehabilitation
- Group B (Active Comparator): Patients in group B recieved cervical traction with 8 kg load combined with standard rehabilitation program. The traction load in this group has an effect on muscular structures of the cervical spine without any actual effect on the remaining anatomical structures (intervertabral disks, joints and ligaments).
  Interventions: Other: Cervical traction; Other: Rehabilitation
- Group C (Experimental): Patients in group C recieved cervical traction with 12 kg load combined with standard rehabilitation program. The traction load in this group has an actual effect on muscles, intervertabral disks, joints, and ligaments of the cervical spine.
  Interventions: Other: Cervical traction; Other: Rehabilitation

INTERVENTIONS:
Other: Cervical traction — Cervical traction procedure was performed using Saunders device. During the procedure, the patient lies in installed in a supine position with 20 degrees of cervical flexion and the physiotherapist gradually increases (5 minutes) the load to the defined kilograms which is maintained for 10 minutes then progressively decreases (5 minutes) the load to zero kilograms. The procedure is performed twice with a rest interval of 5 minutes.
  Other Names: Mechanical intermittent cervical traction
Other: Rehabilitation — The rehabilitation program compiled cervical spine mobilization, stretching of neck muscles and isometric strengthening exercises. Passive stretching of neck muscles groups was carried-out in a seated position with 3 repetition of 30 seconds each. Isometric strengthening exercises of neck extensors were performed in a seated position, against the resistance of the physiotherapist hand for 3 repetitions of 10 seconds each

SUMMARY:
A randomized clinical trial aiming to assess the effect of cervical traction, using different loads, on balance parameters among patients with common cervical radiculopathy.

Authors hypothesized that as cervical traction alleviate radicular pain and improve function it may also improve patient balance parameters. Three different loads of traction are compared Main outcome measures are balance parameters (clinical and stabilometric). Patients are followed for during six months.

DETAILED DESCRIPTION:
A randomized clinical trial was designed to assess the effect of cervical intermittent traction on balance parameters among patients diagnosed with common cervical neuropathy. The diagnosis is confirmed or made by a physical medicine and rehabilitation physician with 15 Y of experience treating musculoskeletal disorders especially cervical neuropathy. Enrolled patients are randomly assigned to one of three groups (A, B and C). Patients are treated with 2 Kg load intermittent cervical traction (A), 8 kg (B) and 12 kg (C). Patients in the three groups are treated additionnally with 12 rehabilitation sessions. Patients are assessed at baseline, at the end of the treatment (1 month), and at 3 and 6 months. Outcomes are mainly clinical balance assessment and stabilometry, and secondary, epidemiological parameters, pain intensity (VAS), cervical spine ROM and proprioception, grip strength, cervical spinal muscle strength, functional status (NDI), the psychological distress (HAD), and Quality of life All parameters are assessed at the Three follow-up points.

ELIGIBILITY:
Inclusion Criteria:

* CR evolving for at least 3 months Well tolerated manual cervical traction test.

Exclusion Criteria:

* Rehabilitation or chiropractic treatment for head or neck pain within the previous 3 months.
* neurological and/or rheumatic diseases involving the cervical spine or which may result in impaired balance.
* Surgery or traumatic damage to the cervical spine.
* Ear, Nose and Throat pathology and ophthalmological disorders causing a balance disorder.
* Diabetes at the stage of neurovegetative complications
* Cardiac arrhythmia
* Neurological impairments (balance disorders, motor and/or sensory deficits).
* Severe osteoporosis or long-term treatment with corticosteroids .

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2023-02-10 (Actual); Primary Completion 2023-06-21 (Actual); Study Completion 2023-12-30 (Actual)

PRIMARY OUTCOMES:
Stabilometric balance assessment 1 | Up to 6 months
  Center of pressure of the foot sway area (Cop/SA) (mm ²)
Stabilometric balance assessment 2 | Up to 6 months
  The lateral displacement length of the center of pressure of the foot (LD) (mm)
Stabilometric balance assessment 3 | Up to 6 months.
  The anteroposterior displacement length of the center of pressure of the foot (AD) (mm)
Stabilometric balance assessment 4 | Up to 6 months
  The lateral displacement velocity (LV) of the center of pressure of the foot (mm/s)
Stabilometric balance assessment 5 | Up to 6 months
  The anteroposterior velocity (AV) of the dispalcement of the center of pressure of the foot(mm/s)
Clinical balance assessment | Up to 6 months.
  For the clinical balance assessment, the Brief-BESTest was used. Six categories included in the test (8 scored):
  1. Biomechanical constraints: Hip strength
  2. Stability limits/verticality: Reach forward
  3. Anticipatory postural responses: Stand on one limb: left and right each scored
  4. Postural responses: Compensatory Stepping right and left each scored
  5. Sensory orientation: Stance on foam with eyes closed
  6. Stability in gait: Get up and Go test Each item is scored: 0 - 3 points (0 representing severe impairment and 3 representing no balance impairment).
  Total score = 24 points (2 items include both a R/L component)

SECONDARY OUTCOMES:
Sociodemographic characteristics 1 | Baseline.
  • Age (years)
Sociodemographic characteristics 2 | Baseline.
  Sex (Male or Female)
Sociodemographic characteristics 3 | Baseline.
  Medical History (Hypertension, diabetes, others)
Sociodemographic characteristics 4 | Baseline.
  Occupation (Employed, unemployed, retired)
Sociodemographic characteristics 5 | Baseline.
  Type of Occupation: Shift work (office work, secretary) or manual labor (heavy manual work, carrying loads)
Sociodemographic characteristics 6 | Baseline.
  Socioeconomic Level: Poor if the salary is below the guaranteed minimum wage (SMIG : around 400 Tunisian Dinars per month) , Average if the salary is between SMIG and three times SMIG, Good if it is more than three times SMIG.
Duration of CR | Baseline.
  The duration of CR is the length of radicular pain evolution in months.
Side of CR | Baseline.
  The side of CR: Right, left, or bilateral
Intensity of CR | Baseline.
  The intensity of radicular pain was assessed using a Visual Analog Scale (VAS) scored out of 100.
• Body Mass Index | Baseline.
  • Body Mass Index (BMI) (kg/m²)
Cervical range of motion (ROM) | Up to 6 months.
  Cervical ROM was measured using the Cervical Range-of-Motion Instrument (CROM; Performance Attainment Associates, St Paul, MN). With its three inclinometers, the CROM device is a useful clinical instrument for measuring the cervical spine's active mobility in flexion, extension, rotation, and lateral flexion.
Cervical proprioception | Up to 6 months.
  Cervical proprioception was assessed using the CROM device. Patient wearing a CROM device is instructed to maintain a neutral head position while sitting (reference position). Patient is asked to close his eyes and move his head passively before returning it to the reference position by the examiner. The angle inaccuracy is measured in degrees by the examiner. The flexion and extension tests are run .
Cervical muscles strength | Up to 6 months.
  Cervical muscles strength was measured using a handheld isometric dynamometer (MicroFET2; Hoggan Health Industries). Measurements were reported in Newton. To assess the strength of the flexor muscles, the dynamometer is placed on the forehead, while for the extensor muscles, it is placed at the back of the head
Handgrip strength (HGS) | Up to 6 months.
  HGS was measured using the Jamar hydraulic handheld dynamometer (Lafayette Instrument Company, USA) and was reported in kilograms.
Neck disability assessment | Up to 6 months.
  The Neck disability index (NDI), a reliable instrument used in clinical practice, was used to assess patients' activities of daily living . It includes 10 items (pain intensity, personal care, lifting, reading, headaches, concentration, work status, driving, sleeping and recreation) each scored from 0 (no disability) to 5 (total disability). The total score is 50 , a higher score indicates a higher disability. The NDI is expressed by percentage. The Arabic version of NDI was delivered to patients.
Psychological status assessment | Up to 6 months.
  The anxiety and depression profiles were assessed using the Hospital Anxiety and Depression scale (HAD). A validated Arabic version of the scale was used. The HAD includes 14 items (7 for anxiety and 7 for depression) rated from 0 to 3 each. The maximum score is 21 for each symptom, and a higher score indicates a poor psychological status . A score less than 7 indicates no depression or anxiety, a score of 8-10 indicates doubtful cases, and a score higher than 11 indicates a certain symptomatology.
Quality of life (QoL) | Up to 6 months.
  The participants' QoL was assessed using the World Health Organization quality of life (WHOQOL-BREF) questionnaire with 4 domains: physical health, psychological, social relationships, and environment. Each domain is reported in percentages, with a higher score indicating better QoL, and a lower score indicating poor QoL.
Kinesiophobia assessment | Baseline.
  The Tampa Scale for Kinesiophobia (TSK) was used to evaluate the kinesiphobia. An Arabic version was administered to patients. The TSK includes 17 items rated from 1 to 4 each, with a total score ranging from 17 to 68. Higher scores reflect greater levels of movement-related fear, and a score higher than 37 indicates the presence of kinesiophobia.

CONTACTS AND LOCATIONS:
Overall Officials: Anis Jellad, Professor, Principal Investigator — University of Monastir, Faculty of Medicine
Locations (1):
- Faculty of Medicine of Monastir, Monastir, Tunisia

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Jellad A, Ben Salah Z, Boudokhane S, Migaou H, Bahri I, Rejeb N. The value of intermittent cervical traction in recent cervical radiculopathy. Ann Phys Rehabil Med. 2009 Nov;52(9):638-52. doi: 10.1016/j.rehab.2009.07.035. Epub 2009 Oct 8. English, French. PMID 19846359
- [Background] Jellad A, Kalai A, Abbes I, Jguirim M, Boudokhane S, Salah Frih ZB, Bedoui MH. The effect of cervical traction on stabilometric parameters in cervical radiculopathy patients: A randomized crossover study. J Back Musculoskelet Rehabil. 2024;37(4):1031-1040. doi: 10.3233/BMR-230270. PMID 38277282